CLINICAL TRIAL: NCT06565000
Title: IMPACT of an Instrumented Measurement on a Performance Assessment in Cerebral Palsy Treatment
Acronym: IMPACT²
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Médico-Chirurgical de Réadaptation des Massues Croix Rouge Française (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: IMPACT²
Record Dates: First submitted 2024-02-06; First posted 2024-08-21 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Cerebral Palsy
Keywords: Quantified Motion Analysis; Performance Assessment; Bimanual Performance; Unilateral Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Experimental)
  Interventions: Other: AHA Not Instrumented then AHA Instrumented
- Group 2 (Experimental)
  Interventions: Other: AHA Instrumented then AHA Not Instrumented

INTERVENTIONS:
Other: AHA Not Instrumented then AHA Instrumented — First, the participant will undergo a performance assessment using the Assisting Hand Assessment test, following the standard protocol in the occupational therapy room. Subsequently, they will proceed to the motion analysis laboratory located across the hall, where an engineer will outfit them with motion capture markers. These markers comprise ultra-reflective spheres affixed to specific anatomical landmarks on their upper limbs using hypoallergenic tape. Afterward, the participant's functional capacity will be evaluated using the Melbourne Assessment. Finally, a second round of assessment using the Assisting Hand Assessment will be conducted.
  Arms: Group 1
Other: AHA Instrumented then AHA Not Instrumented — First, the participant will proceed to the motion analysis laboratory located across the hall, where an engineer will outfit them with motion capture markers. These markers comprise ultra-reflective spheres affixed to specific anatomical landmarks on their upper limbs using hypoallergenic tape. Afterward, the participant's functional capacity will be evaluated using the Melbourne Assessment. Then, will undergo a performance assessment using the Assisting Hand Assessment test.
  Finally, they will go to the occupational therapy room where a second round of assessment using the Assisting Hand Assessment without markers will be conducted.
  Arms: Group 2

SUMMARY:
The goal of this study is to assess the impact of passive reflective markers on bimanual performance assessment scores in children with unilateral cerebral palsy.

The main questions it aims to answer are:

* Is it possible to instrument performance assessment without changing the functionnal behaviour of the patient ?
* How is this behavious modified ?

During their usual occupational therpy assessment at the CMCR Massues, participants will do a second bimanual performance assessment with passive reflection markers taped on their trunk, humerus and forearm.

The glocal scores and sub items scors of both instrumented and non instrumented assessment will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral cerebral palsy
* With an Occupational therapy assessment planed with the duration of the study

Exclusion Criteria:

* Severe cognitive impairment

Ages: 18 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2023-09-18 (Actual); Primary Completion 2024-06-29 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Bimanual Performance Score | 1 day
  The score of the participant at the Assisting Hand Assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- CMCR des Massues, Lyon, France